CLINICAL TRIAL: NCT02298829
Title: Long-term Safety, Curvature Deformity Characterization, and Immunogenicity Over Time in Subjects Previously Treated With AA4500 for Peyronies Disease in Studies AUX-CC-802, AUX-CC-803, AUX-CC-804 and AUX-CC-806
Brief Title: Long-term Safety, Curvature Deformity Characterization, and Immunogenicity Over Time in Subjects Previously Treated With AA4500 for Peyronies Disease
Status: Completed | Type: Observational
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: AUX-CC-810
Record Dates: First submitted 2014-11-20; First posted 2014-11-24 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Peyronie's Disease
Keywords: curvature; bend
MeSH Terms: conditions — Penile Induration; Airway Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for the determination of antibodies to AUX-I and AUX-II and neutralizing antibodies to AUX-I and AUX-II will be collected at each long-term follow-up visit.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No Treatment: Subjects who received AA4500 in a 12-month double blind placebo-controlled study (AUX CC 803 or AUX-CC-804) or in a 9-month open label study (AUX-CC-802 or AUX-CC-806) sponsored by Auxilium Pharmaceuticals, Inc.
  Interventions: Drug: Subjects Previously Treated with AA4500

INTERVENTIONS:
Drug: Subjects Previously Treated with AA4500 — no treatment to be administered - observational only

SUMMARY:
This a Phase 4 non-treatment, long-term follow-up study of subjects who received AA4500 in a 12-month double blind placebo-controlled study (AUX CC 803 or AUX-CC-804) or in a 9-month open label study (AUX-CC-802 or AUX-CC-806) sponsored by Auxilium Pharmaceuticals, Inc. After participation in one of the aforementioned studies, subjects will be followed yearly for up to 4 consecutive long-term follow-up visits with at least 6 months between consecutive visits

DETAILED DESCRIPTION:
At each long-term follow-up visit, subjects will be assessed for adverse events relative to their previous long-term follow-up assessment. Blood samples for the determination of antibodies to AUX-I and AUX-II and neutralizing antibodies to AUX-I and AUX-II will be collected at each long-term follow-up visit.

At each long-term follow-up visit, a flaccid penile examination will be performed and a curvature deformity measurement (with the penis in the erect state) will be recorded. Subjects will also be asked to complete the Peyronie's Disease Questionnaire (PDQ) and the International Index of Erectile Function (IIEF) questionnaire. At each visit, medical, surgical, or other treatments for Peyronie's disease since the last assessment will also be collected and recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Have received at least one injection of AA4500 and completed at least the first or last follow-up visit in one of the Auxilium-sponsored studies (AUX CC-802, AUX-CC-803, AUX-CC-804, or AUX-CC-806).
2. Be able and willing to comply with the follow-up assessments outlined in the protocol, as determined by the investigator.
3. Voluntarily sign and date an informed consent agreement approved by the Institutional Review Board/Independent Ethics Committee (IRB/IEC).

   -

   Exclusion Criteria:

   None

   -

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 750 subjects who received AA4500 and completed at least the first or last follow-up visit in one of the Auxilium-sponsored studies (AUX-CC-802, AUX-CC-803, AUX-CC-804, or AUX-CC-806).
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2014-11; Primary Completion 2018-04-09 (Actual); Study Completion 2018-04-09 (Actual)

PRIMARY OUTCOMES:
To assess the long-term safety of AA4500 in adult men with Peyronies disease | 5 years post treatment

SECONDARY OUTCOMES:
To characterize curvature deformity over time in adult men with Peyronies disease who were treated with AA4500 | 5 years post treatment

OTHER OUTCOMES:
To assess the long-term immunogenicity profile of AA4500 in adult men with Peyronies disease | 5 years post treatment

CONTACTS AND LOCATIONS:
Locations (30):
- United States (30):
  - Alaska Clinical Research Center, LLC, Anchorage, Alaska
  - Urology Assoc Medical Group, Burbank, California
  - South Orange County Med Research Center, Laguna Hills, California
  - San Diego Sexual Medicine, San Diego, California
  - The Urology Center of Colorado, Denver, Colorado
  - South Florida Medical Research, Aventura, Florida
  - Florida Urology Associates, Orlando, Florida
  - Georgis Patsias, M.D., PA, Wellington, Florida
  - Idaho Urologic Institute, Meridian, Idaho
  - Uropartners, LLC, Chicago, Illinois
  - Dupage Medical Group, Winfield, Illinois
  - Urology of Indiana LLC, Avon, Indiana
  - Metropolitan Urology P.S.C, Jefferson, Indiana
  - Kansas City Urology Care, PA, Overland Park, Kansas
  - Chesapeake Urology Research Associates, Glen Burnie, Maryland
  - Chesapeake Urology Research Associates, Towson, Maryland
  - Men's Health Boston, Chestnut Hill, Massachusetts
  - Center for Male Reproductive Medicine, Hackensack, New Jersey
  - Premier Urology Assoc LLC dba AdvanceMed Research, Lawrenceville, New Jersey
  - Community Care Physicians, PC, Albany, New York
  - Bruce R. Gilbert, MD, PhD, PC, Great Neck, New York
  - Manhattan Medical Research Practice PLLC, New York, New York
  - Michael A. Werner, MD PC, Purchase, New York
  - Associated Urologists of North Carolina, Raleigh, North Carolina
  - Tristate Urologic Services dba TUG Research, Cincinnati, Ohio
  - Urologic Consultants of SE PA, Bala-Cynwyd, Pennsylvania
  - Urology Clinics of North Texas, PA, Dallas, Texas
  - Jean Brown Research, Salt Lake City, Utah
  - Virginia Urology, Richmond, Virginia
  - Urology of Virginia, PLLC, Virginia Beach, Virginia